CLINICAL TRIAL: NCT05998174
Title: Faecal Microbiota Transplantation for Microscopic Colitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Sigen Wildt, Consultant, MD, ph.d, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT for MC
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: pilot trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Faecal Microbiota Transplantation — treatment with capsules

SUMMARY:
A pilot study investigating if orally administrated faecal microbiota transplantation capsules have the potential to treat active microscopic colitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of microscopic colitis
* Date of diagnosis/histological confirmation < 12 months
* Active disease according to Hjortswang's criteria

Exclusion Criteria:

* Diagnosed with ulcerative colitis or Crohn's disease
* Diagnosed with celiac disease
* Active gastrointestinal infection
* Previous bowel resection of bowel (except appendectomy)
* Previous cholecystectomy
* Treatment with systemic steroid within 4 weeks, including budesonide
* Antibiotics 3 months prior
* Severe immunodeficiency,
* Pregnancy, planned pregnancy and breastfeeding
* Treatment with constipants such as psyllium, loperamide, bile binders, opium drops or codeine up to 2 weeks before inclusion and during participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Treatment effect | 3 weeks
  Proportion of participants in remission

IPD SHARING:
Plan to Share IPD: No